CLINICAL TRIAL: NCT04737317
Title: Evaluation of Diagnostic Criteria in Cardiac Sarcoidosis - an Observational Study
Brief Title: Diagnostic Criteria in Cardiac Sarcoidosis
Acronym: ELDORADO
Status: Recruiting | Type: Observational
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Borislav Dinov, Head of Ventricular Tachycardia Unit, Heart Center Leipzig - University Hospital
Other Study IDs: 20201231PV1
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Sarcoidosis
MeSH Terms: interventions — Electrocardiography; Caves; Positron Emission Tomography Computed Tomography; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood, serum, myocardial biopsy specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECG, Echo, laboratory tests, CMR, PET-CT, Biopsy — ECG - 12 leads ECG Echo: transthoracic echocardiography laboratory tests: full blood count, electrolytes, creatinine, high sensitive cardiac troponin T, angiontesin converting enzyme, soluble interleukin-2 receptor, cardiac magnetic resonance imaging: 1.5 Tesla scanner, Conventional cine imaging and late gadolinium enhancement imaging PET-CT: 18F-fluorodeoxyglucose (FDG)- positron emission tomograph Biopsy: cardiac biopsy = endomyocardial biopsy, left and right ventricle, at least 5 specimens in formaldehyd and 3 specimens for testing of infectious agents Biopsy: extracardiac biopsy, as accessible according to imaging

SUMMARY:
The purpose of the study is to evaluate the accuracy of the current diagnostic criteria of cardiac sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is an inflammatory condition rarely affecting the heart, exhibiting fluctuating disease activity and eventually leading to ventricular fibrosis. Clinical presentation ranges from no symptoms at all to life-threatening arrhythmias, heart failure and death in severe cases. The heart lesions show patchy distribution and can mimic virtually any other type of cardiomyopathy, which poses significant challenges for the accurate and eary diagnosis.

At present, there are four diagnostic tools and recomendations for diagnosis of cardiac sarcoidosis (CS) that utilize clinical, ECG, laboratory, imaging and biopsy criteria. Recently, it was demonstrated that there is a significant diagreement between these four diagnostic tools. On the other hand, earlier identification of patients with active inflammatory process is necessary, as they are those who will most likely benefit from immunosuppressive therapy.

The aim of this observational study is to evaluate the prognostic significance of the current clinical, ECG, laboratory, imaging and biopsy criteria for diagnosing cardiac sarcoidosis. Patients with suspected cardiac sarcoidosis based on clinical symptoms will recieve elaborate diagnostic work-up consisting of: evaluation of symptoms, family history, occupational hazards, ECG, chest X-ray, laboratory markers for sarcoidosis, positron emission tomography (PET), cardiac magnetic resonance (CMR) as well as endomyocardial biopsy.

In accordance to the recomendations of the current guidelines, the patients will be devided into 3 groups: 1) patients with proven CS; 2) patients with probable CS; and 3) unlikely CS that will serve as a reference group. The patients in first two groups will be treated with immunosuppressive therapy, mainly glucocorticoids (GC). The follow-up at 3, 6, 12 and 24 months will consist of evaluation of the symptoms using dedicated King's Sarcoidosis Questionaire (KSQ), fatigue assessment scale (FAS), Holter-ECG, pacemaker interrogation, laboratory findings, imaging with PET and CMR.

Clinical outcomes will be defined as: 1) improvement of symptoms (FAS score, heart failure class, AV block, ventricular arrhythmias, and KSQ score) and 2) improvement of imaging parameters ( left ventricular ejection fraction, PET activity, myocardial edema, scar in CMR). The outcomes between the groups will be compared using group 3 as reference. Furthermore, patients with improvement with GC (successful therapy) will be compared with those without improvement (unsuccessful therapy) and the predictive value of each diagnostic criterion will be evaluated. Finally, the odds ratios (OR) for each parameter will be used to calculate a diagnostic and predictive score which will be used prospectively to evaluate patients with suspected CS and to guide the therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected CS due to the following presentations:

  1. age < 65 years and new higher degree AV block, causative coronary artery disease excluded
  2. age < 65 years and new ventricular tachycardia, causative coronary artery disease excluded
  3. age < 65 years and ventricular tachycardia, causative coronary artery disease excluded
  4. extracardiac sarcoidosis and cardiac involvement suggested (palpitations, abnormal ECG, abnormal echocardiography)

To diagnose CS one of the following diagnostic tools will be used:

A) World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG)

B) Heart Rhythm Society expert consensus statement on the diagnosis and management of arrhythmias associated with cardiac sarcoidosis

C) Japanese Society of Nuclear Cardiology (JSNC)

Patients whit histological confirmation from myocardial tissue fullfil will be defined as proven CS. (Group 1)

Patients with clinical and imaging findings highly suggesting CS, but without histological confirmation from myocardial biopsy will be defined as probable CS (Group 2)

Patients who do not fullfil the criteria or exhibiting findings suggesting an alternative, more likely diagnosis, will be considered as unlikely CS (Group 3)

Exclusion Criteria:

* unable or unwilling to provide informed consent
* patients who are pregnant or lactating
* noncompliant patients refusing the recommended therapy
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the Heart Center Leipzig, elective and urgent admissions
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical recovery with immunosuppressive therapy | 1 year
  Number of patients showing clinical recovery defined as improvement of at least one of the following: decrease of the heart failure class, decrease of fatigue assessed by FAS score, increase of KSQ score with at least 10 points, reduction of burden of ventricular arrhythmias assessed with Holter ECG or device interrogations, improvement of the AV block
Imaging recovery with immunosuppressive therapy | 1 year
  Number of patients with improvement of the cardiac imaging defined as one of the following: increase of the EF with at least 10%, decrease of the PET activity, decrease of the scar or edema in CMR

SECONDARY OUTCOMES:
Cardiac mortality | 2 years
  Number of patients who died of cardiac reasons
All-cause mortality | 2 years
  Number of patients who died of cardiac or non-cardiac reasons
Unplanned hospitalizations | 2 years
  Number of unplanned hospitalizations due to heart failure or ventricular arrhythmias
Change in LV-EF from baseline | 2 years
  Measured in echocardiography or CMR as at least 10% change of the LV EF, LV EDD
Change in RV function | 2 years
  Measured in echocardiography or CMR as 10% change of RV EF, RV diameter, TAPSE
Patients' quality of life | 2 years
  A dedicated King's Sarcoidosis Questionnaire (KSQ) will be used to assess patients condition. Values from 1 to 100 define the patients' condition with higher scores indicating better condition. Improvement will be defined as increase of the KSQ score with at least 10 points.
VT ablation success | 2 years
  Applies only for patients after VT ablation: Time to VT recurrence
Adverse events of immunosuppressive therapy | 2 years
  Number of patients with significant adverse events related to the immunosuppressive therapy
Changes of immunosuppressive therapy due to lack of success | 2 years
  Number of GC dose increase and/or switch to another medication and/or escalation of therapy adding other immunosuppressive drugs to the GC

CONTACTS AND LOCATIONS:
Overall Officials: Borislav Dinov, MD, Principal Investigator — Heart Center Leipzig - University Hospital, Department Electrophysiology; Laura Ueberham, MD, Study Chair — Heart Center Leipzig - University Hospital, Department Electrophysiology
Locations (1):
- Heart Center of Leipzig, Leipzig, Germany